CLINICAL TRIAL: NCT01371487
Title: An Open-Label, Two-Period, Randomized, Crossover Study to Evaluate the Effect of Food on the Single Dose Pharmacokinetics of the MEK Inhibitor, GSK1120212, in Subjects With Solid Tumors
Brief Title: GSK1120212 Food-effect Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 113709
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): GSK1120212 Dose /Treatment 2.0 mg/Fasted
  Interventions: Drug: GSK1120212
- Treatment B (Experimental): GSK1120212 Dose /Treatment 2.0 mg/high fat, high calorie meal
  Interventions: Drug: GSK1120212

INTERVENTIONS:
Drug: GSK1120212 — Oral/once-daily single doses on Day 1 of Periods 1 and 2

SUMMARY:
The purpose of the this study is to evaluate the effect of a high-fat, high calorie meal on the single dose PK of GSK1120212 in subjects with solid tumors.

DETAILED DESCRIPTION:
open-label, randomized, 2-treatment, 2-period, crossover study with incomplete wash-out to evaluate the effect of a high-fat, high calorie meal on the single dose PK of GSK1120212 in subjects with solid tumors. Subjects will be assigned to a fast/fed sequence according to the randomization code provided to the sites by GSK with subjects randomized to one of 2 possible treatment sequences (Table 1) with each sequence consisting of 2 treatments: a single 2.0 mg dose of GSK1120212 administered under fasted conditions and a single 2.0 mg dose of GSK1120212 administered with a high-fat, high-calorie meal

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria apply:

  1. Male or female; 18 years of age or older at the time of consent
  2. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
  3. Able to swallow and retain oral medication.
  4. Histologically or cytologically confirmed diagnosis of a solid tumor.
  5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Appendix 3).
  6. Adequate baseline organ function defined in Table 5 Definitions for Adequate Baseline Organ Function Absolute neutrophil count greater than or equal to 1.2 × 109/L Hemoglobin greater than or equal to9 g/dL Platelets greater than or equal to 75 × 109/L Prothrombin time (PT), International normalization ratio (INR)a and Partial thromboplastin time (PTT) less than or equal to 1.5 times ULN Hepatic Total bilirubin less than or equal to 1.5 times ULN ALT less than or equal to 2.5 times ULN Renal Creatinine or less than or equal to 1.5 times ULN Calculated creatinine clearance or greater than or equal to 50 mL/min 24-hour urine creatinine clearance greater than or equal to 50 mL/min Cardiac LVEF greater than or equal to LLNc by ECHO or MUGA

     1. INR greater than 1.5 times ULN will be acceptable in case of subjects receiving therapeutic anticoagulants such as warfarin as long as INR is monitored during the study according to clinical practice.
     2. Calculated by the Cockcroft-Gault formula (see Appendix 2).
     3. If LLN is not defined for a given institution, then ejection fraction must be greater than or equal to 50%.
  7. Women of childbearing potential must have a negative serum pregnancy test within 14 days of first dose of study treatment and agree to use effective contraception, as defined in Section 7.1.1, during the study and for 6 weeks following the last dose of study treatment.
  8. Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception as described in Section 7.1.2 from the time of the first dose of study treatment until 16 weeks following the last dose of study treatment (based on the lifecycle of sperm).

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:

  1. Currently receiving cancer therapy (e.g., chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy, or major surgery) within 3 weeks prior to randomization; chemotherapy regimens without delayed toxicity within 2 weeks prior to randomization; or use of an investigational anti-cancer drug within 4 weeks prior to randomization.
  2. Has unresolved Grade 2 or greater toxicity (based on NCI-CTCAE, version 4.0) [NCI Common Terminology Criteria for Adverse Events, 2009] from previous anti-cancer therapy except Grade 2 decreased hemoglobin levels or alopecia.
  3. Has pre-existing peripheral neuropathy of greater than or equal to Grade 2.
  4. Has participated in a clinical trial and has received an investigational product within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product, whichever is longer, prior to the first dose of study treatment in this study.
  5. Has participated in a study that resulted in or made a donation of blood or blood products in excess of 500 mL within 56 days of the first dose of study treatment.
  6. Has presence of active GI disease or other condition (e.g., gastrectomy, bariatric surgery, small or large bowel resection, or cholecystectomy should be excluded) that may interfere significantly with the absorption of drugs. If clarification is needed as to whether a condition will significantly affect absorption of drugs, contact the GSK Medical Monitor.
  7. Has any serious and/or unstable pre-existing medical (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the investigator or GSK Medical Monitor.
  8. Has a history of interstitial lung disease or pneumonitis.
  9. Is currently using a prohibited medication(s) or requires the use of any of the prohibited medications during the study (see Section 8.2).

     • NOTE: Use of anticoagulants such as warfarin is permitted; however, INR must be monitored in accordance with local institutional practice.
  10. Has a history or current evidence/risk of RVO or CSR:

      * History of RVO or CSR, or predisposing factors to RVO or CSR (i.e., uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension or diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes)
      * Visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for RVO or CSR such as:
      * Evidence of new optic disc cupping
      * Intraocular pressure greater than 21 mmHg as measured by tonography
  11. Has symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression

      * Note: Subjects previously treated for these conditions that have had stable central nervous system (CNS) disease (verified with consecutive imaging studies) for greater than 3 months, are asymptomatic and are not currently taking corticosteroids, or are on stable dose of corticosteroids for at least 1 month prior to Day 1 of the study are permitted.
      * Subjects are not permitted to receive enzyme-inducing anti-epileptic drugs (EIAEDs).
  12. Has a QtcB or QTcF (preferred) greater than or equal to 480 msec.
  13. Has a history or evidence of cardiovascular risk including any of the following:
  14. History or evidence of current clinically significant uncontrolled arrhythmias. Exception: Subjects with controlled atrial fibrillation for greater 30 days prior to randomization are eligible.
  15. History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization.
  16. History or evidence of current greater than or equal to Class II congestive heart failure as defined by New York Heart Association (NYHA) (Appendix 4).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05-02 (Actual); Primary Completion 2011-09-30 (Actual); Study Completion 2011-09-30 (Actual)

PRIMARY OUTCOMES:
evaluate the effect of a high-fat, high-calorie meal on the PK of a single dose of GSK1120212 administered to subjects | Predose - 168 hours post dose period 1 and 2
  • Area under the plasma concentration-time curve from time zero (pre-dose) to time t (AUC(0-t)), AUC(0-inf), Cmax, and tmax.

SECONDARY OUTCOMES:
assess the short-term safety and tolerability of single oral doses of 2.0 mg of GSK1120212 administered to subjects | Day 1/periods 1 and 2, Day 8 period 2 and follow-up.
  vital signs, electrocardiograms (ECGs), clinical laboratory tests, and AEs

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, San Antonio, Texas

REFERENCES:
- [Derived] Cox DS, Papadopoulos K, Fang L, Bauman J, LoRusso P, Tolcher A, Patnaik A, Pendry C, Orford K, Ouellet D. Evaluation of the effects of food on the single-dose pharmacokinetics of trametinib, a first-in-class MEK inhibitor, in patients with cancer. J Clin Pharmacol. 2013 Sep;53(9):946-54. doi: 10.1002/jcph.115. Epub 2013 Jul 25. PMID 23893461
- See also: Results for study 113709 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113709?search=study&search_terms=113709#rs